CLINICAL TRIAL: NCT06429046
Title: Effect of Lidocaine Gel and Cold Lidocaine Gel Applied to the Rectal Area on Pain in Patients Who Had Prostate Biopsy With Transrectal Ultrasound: Randomized Controlled Study
Brief Title: Effect of Lidocaine Gel and Cold Lidocaine Gel on Pain in Patients Who Had Prostate Biopsy With Transrectal Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Sevda Fırat, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CukurovaUSFırat2
Record Dates: First submitted 2024-05-09; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer XXX; TRANSRECTAL ULTRASOUND-GUIDED PROSTATE BIOPSY
Keywords: Cold application

STUDY DESIGN:
Intervention Model Description: This study was planned to compare the effects of lidocaine gel and cold lidocaine gel application to the rectal area on the pain level in patients who underwent TRUSG-guided prostate biopsy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CONTROL (No Intervention): For patients in the control group, "Personal Information Form" will be applied before the procedure and pain will be evaluated with "Numeric Pain Scale".
  NPS will be applied at the beginning of the procedure when the ultrasound probe is placed (NPS-1), 5 minutes after the procedure (NPS-2) and at the end of the procedure when the probe is removed (NPS-3).
  However, no treatment will be performed on control group patients.
- LIDOCAINE GEL (LG) (Experimental): Data will be collected in two stages. To LG group patients, 20 ml lidocaine gel will be applied intrarectally (double application: 5cc to the perianal region, covering the anal sphincter, the remaining 15cc into the rectum) 5 minutes before the transrectal ultrasound probe is placed in the rectum. Patients in the LG group will be administered a "Personal Information Form" before the procedure, and their pain will be evaluated with the "Numeric Pain Scale". NPS will be applied at the beginning of the procedure when the ultrasound probe is placed (NPS-1), 5 minutes after the procedure (NPS-2) and at the end of the procedure when the probe is removed (NPS-3).
  Interventions: Other: LIDOCAINE GEL
- COLD LIDOCAINE GEL (CLG) (Experimental): Similarly, patients in the CLG group will be administered "Personal Information Form" before the procedure and pain will be evaluated with "Numeric Pain Scale". In CLG group patients, 20 ml of cold lidocaine gel kept in the refrigerator at +4 0C will be applied intrarectally (double application: 5cc to the perianal region, including the anal sphincter, the remaining 15cc into the rectum) 5 minutes before the transrectal ultrasound probe is placed into the rectum.NPS will be applied at the beginning of the procedure when the ultrasound probe is placed (NPS-1), 5 minutes after the procedure (NPS-2) and at the end of the procedure when the probe is removed (NPS-3).
  Interventions: Other: COLD LIDOCAINE GEL

INTERVENTIONS:
Other: LIDOCAINE GEL — To LG group patients, 20 ml lidocaine gel will be applied intrarectally (double application: 5cc to the perianal region, covering the anal sphincter, the remaining 15cc into the rectum) 5 minutes before the transrectal ultrasound probe is placed in the rectum.
  Arms: LIDOCAINE GEL (LG)
Other: COLD LIDOCAINE GEL — In CLG group patients, 20 ml of cold lidocaine gel kept in the refrigerator at +4 0C will be applied intrarectally (double application: 5cc to the perianal region, including the anal sphincter, the remaining 15cc into the rectum) 5 minutes before the transrectal ultrasound probe is placed into the rectum.
  Arms: COLD LIDOCAINE GEL (CLG)

SUMMARY:
Prostate cancer is one of the most common types of malignancy in men. Transrectal ultrasound-guided prostate biopsy (TRUSG-PBx) is considered the current gold standard method in the diagnosis of prostate cancer. Some patients experience serious discomfort during the procedure because the ultrasound probe is placed in the rectal area. Although no anesthetic or analgesic is used in some centers during the prostate biopsy procedure, in some centers lidocaine gel, cream or spray is applied before entering the rectal area, and lidocaine ampoule is injected during the procedure. However, most patients experience pain and discomfort due to the way the procedure is performed.

Today, in addition to pharmacological methods, non-pharmacological methods are also used to control pain. Cold application has an important place among non-pharmacological methods. In this randomized controlled intervention study, the effect of cold lidocaine gel application on pain level in patients undergoing transrectal ultrasound-guided prostate biopsy (TRUSG-PBx) will be evaluated. In this study, it is thought that application of cold lidocaine gel will reduce the pain level of patients.

The research will be conducted at the Urology Polyclinic of Çukurova University Faculty of Medicine Balcalı Practice and Research Hospital. The sample of the research; Ç.Ü.T.F. Volunteer patients who have undergone prostate biopsy at the Urology Polyclinic of Balcalı Practice and Research Hospital and meet the research criteria will be recruited. Patients consisting of 3 groups: control, experiment 1 (Lidocaine Gel) and experiment 2 (Cold Lidocaine Gel) will be determined by randomization. A power analysis was carried out by obtaining statistical support for the sample size. As a result of the sample calculation calculated with power with a confidence interval of 95%, beta value of 95% and alpha value of 0.05, a total of 114 patients will be included, 38 each in the control group, Lidocaine gel and Cold Lidocaine Gel groups. . Data will be collected with the "Personal Information Form" and "Pain Assessment Form". The data will be analyzed in the SPSS (Statistical Package for the Social Sciences) package program.

In this context, in our study, the effect of lidocaine gel and cold lidocaine gel applied to the rectal area on the pain level in patients who underwent transrectal ultrasound-guided prostate biopsy will be evaluated and the effect of cold application on pain control will be compared. This result will make great contributions to patient benefit in terms of pain management.

DETAILED DESCRIPTION:
Prostate cancer is one of the most common types of malignancy in men. According to GLOBOCAN (Global cancer statistics) 2020 data, the age-standardized incidence rate of prostate cancer varies between 11.3-37.5 per hundred thousand in the world, depending on the development level of the countries, and it is seen to be 42.5 per hundred thousand in our country. It ranks second after lung cancer in terms of incidence in men in our country and in the world. Prostate cancer screening aims to reduce mortality and morbidity by detecting prostate cancer at an early stage. Digital rectal examination (DRE), prostate specific antigen (PSA) value, transrectal ultrasonography (TRUS) and biopsy are used to diagnose prostate cancer. Ultrasound-guided prostate biopsy has been used since 1981 and is one of the most important urological diagnostic methods. Transrectal ultrasound-guided prostate biopsy (TRUSG-PBx) is currently considered the gold standard method in the diagnosis of prostate cancer. In the TRUSG-guided biopsy procedure, after the patients are placed in the left lateral or lithotomy position, the needle-guided rectal probe is inserted into the anal canal with the help of lubricating gel, and the prostate tissue is monitored under USG guidance and a biopsy is taken. The procedure takes approximately 20 minutes, and approximately 15 minutes pass during the entry and exit of the probe into the rectal area. In recent years, the importance of pain control has increased due to prostate biopsy being performed on younger patients, biopsies being taken from more quadrants, and repeated prostate biopsies. Due to severe pain, the rate of tolerance of the procedure by the patient decreases, and this may lead to a decrease in the number of biopsy samples taken from the planned quadrant and a decrease in cancer detection rates. Therefore, ensuring pain control and increasing patient tolerance in TRUSG-PBx is extremely important. Many different methods are used to reduce pain and discomfort. In recent studies, local anesthesia is used in transrectal ultrasound-guided prostate biopsies; Methods such as periprostatic nerve block (PPSB), lidocaine injection, intrarectal lidocaine gel, transperineal periprostatic block (TPPB with gel combination), low-dose spinal anesthesia and intravenous (IV) sedation application have been used and results have been reported showing that these methods increase the pain tolerance in the patient. One of the most important obstacles to the biopsy process is anal area pain. The pain felt during the biopsy occurs for 2 reasons:

1. Pain felt when the biopsy needle penetrates the prostate capsule and enters the stroma.
2. Pain caused by stretching of the anal sphincter as the transrectal ultrasound probe enters the anus (passing the ultrasound probe through the anus, advancing it into the rectum, and manipulating it within the rectum).

For periprostatic nerve blockade before biopsy, penetration into the rectum with a rectal probe is required before anesthesia, and this first penetration is the main cause of the patients' complaints. Due to pain resulting from anal canal sensation during biopsy, intrarectal local anesthesia, which is highly absorbed through the rectal mucosa, is frequently used. Although the procedure is easy to perform and causes very low mortality, efforts to reduce the discomfort and pain that patients may feel lead to the development of new protocols for pre-procedure preparations and anesthesia and analgesia. Most patients who will undergo transrectal biopsy experience anxiety due to the possibility of the result being cancer, the psychological discomfort caused by the fact that the procedure will be performed rectally, and the procedure is painful for the patient. Nurses have an important and indispensable role in pain control and within the team. To reduce pain, nurses; They should inform patients about pain preventive approaches and pain control methods and give the message to patients that everything necessary has been done before painful procedures. Nurses should also apply non-pharmacological methods to reduce the consumption of analgesic drugs or increase their effect by providing adequate analgesia. The patient, whose anxiety decreases, will perceive the intensity and duration of pain as decreased as his sense of pain control will improve.

Non-pharmacological methods are used alone or together with pharmacological methods in order to reduce the use of analgesics and at the same time improve the quality of life of the patient by relieving the patient's pain as much as possible. Cold application also has an important place among non-pharmacological methods.

Cold application is effective in reducing pain, indirectly or directly. It indirectly reduces pain by eliminating edema, swelling and muscle spasm resulting from inflammation or trauma, and has a direct effect by changing the conduction properties of peripheral nerves. In this context, evidence-based studies should be examined and pharmacological and non-pharmacological methods that reduce pain should be used in patient care areas.

A study in the literature showed that applying intrarectal lidocaine gel by massaging the anal area increases patient tolerance and provides balanced and adequate anesthesia at every stage of the biopsy.

In another study in the literature, they compared the application of three intrarectal anesthesia methods along with periprostatic nerve block (periprostatic nerve block with intrarectal lidocaine gel, lidocaine cream and indomethacin suppository) during transrectal ultrasonography-guided prostate biopsy. They stated that intrarectal lidocaine cream application together with PPSB provided more effective pain control.

In the literature, studies conducted to evaluate the effect of cold application on pain during removal of mediastinal and thorax tubes have observed that the application reduces pain, and it has been stated that applying cold to the entry point of the chest tubes reduces the pain and the amount of analgesic consumption during movement and coughing.

As can be seen, various studies have been conducted to determine which anesthesia technique will reduce pain and to evaluate the rectal pain and sensitivity caused by the probe. However, it is still controversial which local anesthesia method is more suitable and will cause less pain. However, although there are many national and international studies on the subject in the literature, no experimental study has been found on the effect of cold lidocaine gel application on the pain level in patients who underwent transrectal ultrasound-guided prostate biopsy. The purpose of our research, which we planned in the light of this information, is to compare the effect of applying cold lidocaine gel to the rectal area on the pain level in patients who underwent transrectal ultrasound-guided prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Being able to communicate effectively,
* Being over 40 years old,
* Being literate,
* Volunteering to participate in the research.

Exclusion Criteria:

* Having a previous history of chronic pain,
* Having alcohol and drug addiction,
* Having bleeding diathesis and active urinary tract infection,
* Having a cognitive disorder, neurological or psychiatric disease,
* Having a disease in the anal and rectal area (wound, fistula, fissure, hemorrhoids, etc.).
* Not agreeing to participate in the research.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — PROSTATE
Enrollment: 120 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Pain Evaluation Form | The first 24 hours: NPS 1, 2, 3.
  The scale used in the first part of this form, which aims to evaluate pain severity, is the Numerical Pain Scale (NPS). On this scale, it starts with no pain (0) and reaches the level of unbearable pain (10). It was applied according to the determined measurement times of the patients [At the beginning of the biopsy/while the ultrasound probe was being inserted (NPS) -1), During the biopsy/5 minutes after the ultrasound probe was placed (NPS-2), At the end of the biopsy/when the ultrasound probe was being removed (NPS-3)].

SECONDARY OUTCOMES:
Personal Information Form | Personal Information Form was applied before the transaction
  This form, prepared by the researchers in line with the literature, aims to determine the individual characteristics of the patients (age, marital status, height/weight/body mass index, educational status, chronic disease status, previous rectal examination/procedure/biopsy, previous rectal 8 questions are included (e.g. pain status and level experienced during the examination/procedure/biopsy performed in the area).

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Sariçam, Turkey (Türkiye)